CLINICAL TRIAL: NCT02588651
Title: A Phase II Study of Single Agent Brentuximab Vedotin in Relapsed/Refractory CD30 Low (<10%) Mature T Cell Lymphoma (TCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deepa Jagadeesh (Other)
Responsible Party: Sponsor-Investigator, Deepa Jagadeesh, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1415
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: T-cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Hepato-splenic T-cell Lymphoma; Adult T-cell Leukemia/Lymphoma; Enteropathy Associated T-cell Lymphoma; NK T-cell Lymphoma
Keywords: Lymphoma; Leukemia; Brentuximab Vedotin
MeSH Terms: conditions — Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Enteropathy-Associated T-Cell Lymphoma; Lymphoma, Extranodal NK-T-Cell; Lymphoma; Leukemia | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab vedotin (Experimental): Brentuximab vedotin 1.8 mg/kg intravenously (IV) once every 3 weeks
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — study drug given intravenously to determine efficacy in study diseases

SUMMARY:
This study will include patients with mature T-cell lymphoma (MTCL) that has been treated with at least one type of chemotherapy, but is not responding or coming back after the previous treatment.

This clinical trial uses a drug called Brentuximab Vedotin. The Food and Drug Administration (FDA) has approved Brentuximab Vedotin for sale in the United States for certain diseases. Brentuximab is still being studied in clinical trials like this one to learn more about what its side effects are and whether or not it is effective in the disease or condition being studied.

Brentuximab Vedotin is a type of drug called an antibody drug conjugate (ADC). ADCs usually have 2 parts; a part that targets cancer cells (the antibody) and a cell killing part (the chemotherapy). Antibodies are proteins that are part of your immune system. They can stick to and attack specific targets on cells. The antibody part of Brentuximab Vedotin sticks to a target called CD30. CD30 is an important molecule on some cancer cells (including non Hodgkin lymphoma) and some normal cells of the immune system. The cell killing part of Brentuximab Vedotin is a chemotherapy called monomethyl auristatin E (MMAE). It can kill cells that the antibody part of Brentuximab Vedotin sticks to. Brentuximab Vedotin has also been shown to kill cancer cells with levels of CD30 that cannot be seen by traditional methods.

This study is being done to test if the study drug has an effect on Mature T cell Lymphoma with such low levels of a target called CD30 and how your disease respond to the study drug.

DETAILED DESCRIPTION:
Primary Objective

• To determine overall response rate (CR+PR) of brentuximab vedotin in CD30 low (<10%) relapsed or refractory T cell lymphoma (TCL)

Secondary Objective(s)

* Complete remission (CR) rate
* Duration of response (DOR)
* Progression free survival (PFS)
* Overall survival (OS)
* Time to treatment failure (TTF)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed/refractory CD30 low (<10%) TCL: including peripheral TCL not otherwise specified (PTCL NOS), angioimmunoblastic T cell lymphoma (AITL), hepato-splenic T cell lymphoma (HTCL), adult T cell leukemia/lymphoma (ATLL), enteropathy associated T cell lymphoma (EATL), adult T cell leukemia/lymphoma (ATLL), enteropathy associated T cell lymphoma (EATL), NK T cell lymphoma (NK/TCL)
* At least 1 prior chemotherapy regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. ECOG Performance Status (PS) 3 will be permitted if the decreased PS is attributed to the lymphoma
* Adequate organ function

  * Bilirubin ≤1.5X upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3X ULN even in patients with documented hepatic involvement with lymphoma
  * Serum creatinine clearance ≥30 ml/min
  * Absolute neutrophil count (ANC) ≥1000/μL (unless documented bone marrow involvement with lymphoma)
  * Platelet count ≥50,000/μL (unless documented bone marrow involvement with lymphoma)
* At least 6 weeks from autologous stem cell transplantation
* At least 3 months from allogeneic stem cell transplantation and off immunosuppression and no evidence of graft versus host disease (GVHD)
* Previous treatment with brentuximab vedotin will be allowed if it was done 6 months prior to enrollment and patient was not refractory
* Measurable disease ≥1.5 cm seen on computed tomography (CT) scan and Fluorodeoxyglucose (FDG) avid disease on positron emission Tomography (PET) scan. Splenomegaly measuring >12 cm, if attributed to TCL and/or positive bone marrow involvement with lymphoma are also eligible.
* Females of childbearing potential must have a negative serum or urine pregnancy test result within 7 days prior to the first dose of study treatment. Women of child-bearing age must agree to use an effective contraception method during the study and for at least 6 months following the last dose of study drug.
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of study drug.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Anaplastic large cell lymphoma (ALCL) both alk positive and negative
* Cutaneous T cell lymphomas except transformed Mycosis fungoides (MF)
* Prior treatment with Brentuximab in the last 6 months or previously refractory to Brentuximab Vedotin (BV) or had progressive disease (PD) while on BV
* Pregnancy or breast feeding women
* Prior malignancy within the past 3 years except non melanoma skin cancer or other localized cancer treated with curative intent
* Presence of grade >2 peripheral neuropathy or patients with the demyelinating form of Charcot-Marie-Tooth syndrome.
* Presence of central nervous system (CNS) involvement requiring active treatment
* History of progressive multifocal leukoencephalopathy (PML)
* Myocardial infarction within the past 6 months
* Patients with the following medical conditions that could affect their participation in the study:

  * any active acute or chronic or uncontrolled infection
  * liver disease including history of viral hepatitis B or C, evidence of cirrhosis, chronic active or persistent hepatitis
  * a known history of HIV
  * symptomatic cardiac disease, including congestive heart failure, coronary artery disease, and arrhythmias
* Prior hypersensitivity to any component in the ADC formulation
* Treatment with chemotherapy or investigational agents within 2 weeks of start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Jagadeesh, MD, MPH, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Paolo Caimi, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Wayne State University, Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brentuximab Vedotin
Started | 23
Completed | 2
Not Completed | 21
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1
Not completed — Lack of Efficacy | 13
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 23
Age, Customized [Number; unit: years]
  20-29 | 3
  40-49 | 2
  50-59 | 3
  60-69 | 9
  70-79 | 4
  Unknown | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary objective is to evaluate overall response rate (ORR). Overall response rate will be estimated by the total number of patients who achieve a CR and PR divided by the total number of patients who received treatment. Response was assessed using CT scans according to the revised Cheson criteria.
  * CR is defined as complete resolution of all clinically detectable disease and disease related symptoms that were present prior to therapy
  * PR is defined as at least 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses Patients should have completed at least 1 cycle of treatment to be evaluable for ORR.
Time Frame: Three years after end of treatment, up to 49 months
Population: 1 participant did not complete one cycle; 3 additional participants did not have response data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 19
percentage of participants | 89.5 [75.5 to 100]

2. Secondary Outcome: Complete Response
Description: Complete Response is defined as complete resolution of all clinically detectable disease and disease related symptoms that were present prior to therapy. A post-treatment residual mass of any size is permitted as long as it is PET negative. CR rate was calculated by dividing the total number of patients who have achieved a complete response by the total number of patients who received treatment.
Time Frame: Three years after end of treatment, up to 49 months
Population: 1 participant did not complete one cycle; 3 additional participants did not have response data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 19
percentage of participants | 10.5 [0 to 24.3]

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from treatment initiation into the study to disease progression or death due to any cause. The distribution of PFS will be estimated using the Kaplan-Meier method. Disease progression may be defined as the date of documentation of a new lesion or enlargement of a previous lesion, or the date of the scheduled clinic visit immediately after radiologic assessment has been completed. For a patient who is alive without progression at the end of study follow-up, observation of PFS is censored on the date of last contact.
Time Frame: Three years after end of treatment, up to 49 months
Population: 1 participant did not have at least one dose
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 22
Month | 8.0 [5.3 to 12.3]

4. Secondary Outcome: Overall Survival
Description: The overall survival (OS) is defined as the time from treatment initiation to the time of death due to any cause. For a patient who is alive at the end of study follow-up, observation of OS is censored on the date of last contact. The distribution of OS will be estimated using the Kaplan-Meier method.
Time Frame: Three years after end of treatment, up to 49 months
Population: 1 participant did not have at least one dose
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 22
Month | 10.8 [5.6 to 20.8]

5. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) among responders is defined as the time from first documentation of objective tumor response (CR or PR) to the time of first progression or death due to any cause.
Time Frame: Three years after end of treatment, up to 49 months
Population: 6 participants did not have ORR
Measure: Median (Inter-Quartile Range); unit: Month
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 17
Month | 5.4 [2.8 to 17.6]

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to treatment failure (TTF) is defined as the time from treatment initiation to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death. Date of last follow-up was collected for patients who did not have disease progression, but it is unknown for which reasons treatment was stopped for these patients. In this case, time to treatment failure (TTF) is the same as time to progression.
Time Frame: Up to 13 months after start of treatment
Population: 6 participants did not have progression at last follow-up
Measure: Median (Inter-Quartile Range); unit: Month
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 17
Month | 7.4 [5.1 to 12.1]

7. Secondary Outcome: Time to Response (TTR)
Description: Time to treatment failure (TTR) is defined as time from treatment initiation to first documentation of objective tumor response (CR or PR).
Time Frame: Three years after end of treatment, up to 49 months
Population: 6 participants did not have ORR
Measure: Median (Inter-Quartile Range); unit: Month
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 17
Month | 2.7 [2.5 to 2.7]

ADVERSE EVENTS:
Time Frame: All AEs (regardless of relationship to study drug) captured from the time the subject signs the ICF through the end of the safety-reporting period, approximately 4 years.
Arm/Group | Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 17/23
Serious Adverse Events (participants affected / at risk) | 10/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin (N=23)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Capillary leak syndrome (Vascular disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fever (General disorders) | 4 (8)
Fatigue (General disorders) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) — Melena
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Infections and infestations - Other, specify - (Investigations) | 1 (1) — bacteremia
Kidney infection (Renal and urinary disorders) | 1 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin (N=23)
Abdominal pain (Gastrointestinal disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 7
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Capillary leak syndrome (Vascular disorders) | 1
Chills (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 6
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema face (General disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 10
Fever (General disorders) | 8
Flu like symptoms (General disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — tongue lesion
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Edema (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Genital edema (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Pain Bilateral Hips
Headache (Nervous system disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Nail infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Blood and lymphatic system disorders) | 6
Papulopustular rash (Infections and infestations) | 1
Paresthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 9
Presyncope (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Bronchitis
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Rhinitis
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 1 — C. Difficile infection
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 4
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — lipomas
Tinnitus (Ear and labyrinth disorders) | 1
Thrush (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
White blood cell decreased (Investigations) | 2
Weight loss (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT02588651/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT02588651/ICF_001.pdf